CLINICAL TRIAL: NCT03078114
Title: Central Mechanism of Manual Therapy for Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Chiropractic Mutual Insurance Company Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12919
Record Dates: First submitted 2017-03-01; First posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal Manipulation (Experimental): Subjects with subacute low back pain. Subjects will receive 6 treatments of Spinal Manipulation (SM) over 2 consecutive weeks
  Interventions: Other: Spinal Manipulation
- Placebo Spinal Manipulation (Placebo Comparator): Subjects with subacute low back pain. Subjects will be asked to visit the clinic for 6 times. The clinician will go through SM motions but the spine will not actually be manipulated.
  Interventions: Other: Placebo Spinal Manipulation

INTERVENTIONS:
Other: Spinal Manipulation — The subject will be asked to lay down and bend in a specific way. The clinician will apply force to certain areas to manipulate the spine.
  Arms: Spinal Manipulation
Other: Placebo Spinal Manipulation — The subject will be asked to lay down and bend in a specific way. The clinician will apply force to certain areas to simulate manipulating the spine.
  Arms: Placebo Spinal Manipulation

SUMMARY:
The purpose of this study is to examine the change of nervous system activity before and after spinal manipulation treatment program in people with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subacute low back pain
* Ability to read and understand English

Exclusion Criteria:

* Previous low back surgery
* Severe structural spinal deformity
* Neurological compromise resulting in current nerve root entrapment
* Spinal cord compression
* Tumor
* Severe spinal instability
* Severe osteoporosis
* Psychiatric disease
* Head trauma
* Spinal infection
* Known cardiovascular or metabolic disease
* Known neurological, neuromuscular or orthopedic problems that might prevent them from participating in manual therapy interventions
* Pregnancy
* Mini-Mental State Examination score < 25
* Body Mass Index (BMI) < 18 or > 30
* Pain or paresthesia below the knees
* Systemic illness known to affect sensation i.e. diabetes
* Acute and/or chronic pain condition unrelated to LBP

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2012-05; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Pain Threshold measured using Pain Pressure Threshold (PPT) testing | Change from Pre-treatment to Post-treatment, 2 Weeks
  Outcome will be measured using Pain Pressure Threshold (PPT) testing. Pressure will be applied to subjects using a digital algometer. Three trials for PPT will be done and the mean value will be calculated.

SECONDARY OUTCOMES:
Change in function measured using the Oswestry Disability Index (ODI) | Change from Baseline to Week 2
  Outcome will be measured using the Oswestry Disability Index (ODI). Subjects answer to questions. Their responses indicate no impact to great impact. Scores for each question range from 0 to 5. Total score for the ODI is 50. The higher the score, the greater level of disability/function.
Change in Low Back Pain measured using the Numerical Pain Rating Scale (NPRS) | Change from Baseline to Week 2
  Outcome will be measured using the Numerical Pain Rating Scale (NPRS). Pain intensity will be assessed using an 11-point scale. Scores on the scale range from "0" indicating no pain, "1" slight pain, and "10" strongest imaginable pain.
Change in Fear Avoidance Beliefs Questionnaire (FABQ) | Change from Baseline to Week 2
  The FABQ is completed by the subject. It determines the level of fear and avoidance about work and physical activity. The measure is comprised of two subscales: a four item physical activity subscale (FABQ-W), and a seven-item work subscale (FABQ-W). An elevated FABQ score is predictive of the development of chronic disability in low back pain (LBP) patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Liu, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University Of Kansas Medical Center, Kansas City, Kansas
  - University of Saint Mary, Leavenworth, Kansas

REFERENCES:
- [Derived] Bond BM, Kinslow CD, Yoder AW, Liu W. Effect of spinal manipulative therapy on mechanical pain sensitivity in patients with chronic nonspecific low back pain: a pilot randomized, controlled trial. J Man Manip Ther. 2020 Feb;28(1):15-27. doi: 10.1080/10669817.2019.1572986. Epub 2019 Mar 5. PMID 30935324